CLINICAL TRIAL: NCT00579878
Title: Triple III Comparison of Leflunomide Alone Versus Two DMARD Combinations (Leflunomide-Hydroxychloroquine-Sulfasalazine or Methotrexate-Hydroxychloroquine-Sulfasalazine) in the Treatment of Rheumatoid Arthritis
Brief Title: Triple III Comparison of Leflunomide Alone Versus Two DMARD Combinations in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0012-01-FB
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Leflunomide; Methotrexate; Sulfasalazine; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Leflunomide alone vs combination therapy (Active Comparator): Group A: Leflunomide alone
  Interventions: Drug: Leflunomide
- Methotrexate-Sulfasalazine-Hydroxychloroquine (Active Comparator): Methotrexate, Sulfasalazine, Hydroxychloroquine.
  Interventions: Drug: Methotrexate-Sulfasalazine-Hydroxychloroquine
- Leflunomide-Sulfasalazine-Hydroxychloroquine (Active Comparator): Leflunomide-Sulfasalazine-Hydroxychloroquine
  Interventions: Drug: Leflunomide-Sulfasalazine-Hydroxychloroquine

INTERVENTIONS:
Drug: Leflunomide — A loading dose of 100 mg (or placebo) for three (3) days will be given. Following that three-day period, a dose of 20 mg/day will be maintained throughout the remainder of the study. This dose may be decreased to 10 mg/day at the discretion of the treating physician if minor toxicities occur (e.g., diarrhea, liver enzyme elevations
  Other Names: Arava®
  Arms: Leflunomide alone vs combination therapy
Drug: Methotrexate-Sulfasalazine-Hydroxychloroquine — Methotrexate:
  dosing starts at 10mg/week (4 tabs/wk). If total remission (according to ACR criteria found in Appendix II) has not been achieved and the labs are acceptable at the 8-week evaluation, the dose increased to 15 mg/week (6 tabs/wk);at the 16-week evaluation, the dose increased to 20 mg/week (8 tabs/wk). This dose will remain stable until the end of the study.
  Sulfasalazine: dosing will start at 500 mg bid (1000 mg/day). This dose will remain steady until the 24-week evaluation. If total remission has not been achieved by this time and the labs remain acceptable,dose will be increased to 1000 mg bid (2000 mg/day) Hydroxychloroquine: dosing will be started and maintained throughout the study at 200 mg bid (400 mg/day).
  Other Names: Trexall, Rheumatrex; Azulfidine®; Plaquenil®
  Arms: Methotrexate-Sulfasalazine-Hydroxychloroquine
Drug: Leflunomide-Sulfasalazine-Hydroxychloroquine — Leflunomide: dose of 100 mg (or placebo) for three (3) days. Followed by a dose of 20 mg/day will be maintained throughout the remainder of the study. dose may be decreased to 10 mg/day at the discretion of the treating physician if minor toxicities occur Sulfasalazine: dosing will start at 500 mg bid (1000 mg/day). This dose will remain steady until the 24-week evaluation. If total remission has not been achieved by this time and the labs remain acceptable, dose will be increased to 1000 mg bid (2000 mg/day) Hydroxychloroquine: dosing will be started and maintained throughout the study at 200 mg bid (400 mg/day).
  Other Names: Arava®; Azulfidine®; Plaquenil®
  Arms: Leflunomide-Sulfasalazine-Hydroxychloroquine

SUMMARY:
The study has been designed as a 48-week, double-blind, randomized, controlled study comparing the use of leflunomide alone to combinations of leflunomide-sulfasalazine-HCQ, and methotrexate-sulfasalazine-HCQ.

DETAILED DESCRIPTION:
Objectives: The combination of methotrexate-sulfasalazine-hydroxychloroquine has been shown to be more effective than methotrexate alone or the double combination of methotrexate-sulfasalazine or methotrexate-hydroxychloroquine. The objective of this study is to look at the safety and efficacy of a new DMARD, leflunomide, alone or in combination with traditional DMARDs (sulfasalazine and hydroxychloroquine).

Research Design: This protocol has been designed as a 48 week, double blind, randomized, prospective and controlled. A total of 180 subjects will be enrolled, and randomly assigned to one of three study arms (60 subjects in each arm): 1) leflunomide alone; 2) leflunomide-sulfasalazine-hydroxychloroquine; 3) methotrexate-sulfasalazine-hydroxychloroquine. All subjects will receive an identical number of medications in a combination of active drug and placebo. Patients are further stratified into two groups: methotrexate-naïve (no history of methotrexate); and methotrexate-failure (failed to achieve clinical response at top dose of 20 mg/week for at least 8 weeks). Methotrexate-naïve patients will start the study at 10 mg/week methotrexate with possible increases at next evaluations dependent on remission criteria. Methotrexate-failure patients will start the study at the top study dose of 20 mg/week and remain at that dose for the entire study.

Methodology: All patients will be recruited from outpatient academic, private practice, and VA rheumatology clinics. Subjects will be between the ages of 19 and 80 years. No pediatric subjects will be enrolled. No enrollment restrictions are based on race, ethnic origin or gender. Inclusion criteria includes: formal diagnosis of rheumatoid arthritis per ACR criteria; disease duration of >6 months; at least 6 swollen and 6 tender joints on examination; and negative urine pregnancy test for premenopausal females. Specific exclusion criteria includes: previous treatment with leflunomide or combination DMARDs; abnormal lab values; history of allergy to sulfa, aspirin or tartrazine; any significant comorbid diseases; and unwillingness to avoid alcohol. Study subjects will return for evaluations every 8 weeks. All patients will be monitored for efficacy and signs of drug toxicity throughout the study by laboratory examination (CBC with platelets, AST or ALT, albumin, creatinine, and erythrocyte sedimentation rate), hand x-rays, retinal examination, and chest x-rays (if indicated). Every six months subjects will be asked to complete the ClinHAQ and SF36 questionnaires, designed to evaluate the effect of RA on daily live (ADLs). Subjects will be withdrawn from the study: due to pregnancy; serious adverse event not alleviated by symptomatic treatment; recurrent toxicity that reappears after treatment or drug suspension; lack of efficacy (20% improvement by week 32); non-compliance with the protocol; or withdrawal of consent. The primary study outcome measures were planned before data collection began.

Clinical Relationship: Rheumatoid arthritis is a chronic disease affecting a large proportion of the population. It produces significant morbidity and may result in premature mortality. The majority of patients with RA remain on disease-modifying agents for less than two years because of toxicity or lack of efficacy. Because of the failure of standard therapies to consistently halt and slow the progression of disease and the incidence of side effects, new approaches are clearly needed.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or 19 years and less than or 80 years old
* Duration of disease greater or equal to 6 months
* Diagnosis of RA with criteria
* Negative urine pregnancy test
* Be capable of understanding and giving written, voluntary informed consent
* Must present with at least six swollen and six tender joints at the screening evaluation

Exclusion Criteria:

* Patients treated previously with leflunomide
* Patients that have been treated with methotrexate in combination with any of the study drugs
* Patients with a history of allergy to, or any history of significant clinical or laboratory adverse experience associated with any of the study drugs
* Doses of oral steroids that are either unstable or greater than 10mg/day
* Stage IV disease or other significant disease including chest x-rays that show evidence of rheumatoid lung disease. Stage IV disease is defined as x-ray evidence of cartilage/bone destruction with fibrous or bony ankylosis; creatinine greater than 2.0mg/dL, AST or ALT greater normal
* Any significant liver, renal , hematologic, pulmonary, cardiovascular disease (including uncontrolled hypertension), any active peptic ulcer disease, or visual problems including a recent decrease in acuity, retinal disease, or macular degeneration
* Patients who are not willing to abstain from alcohol consumption
* Women of childbearing potential who are not practicing a successful method of contraception, or wish to become pregnant
* Patients that are unable to understand the study procedures and/or give written informed consent.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2001-03-27 (Actual); Primary Completion 2010-03-11 (Actual); Study Completion 2010-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R O'Dell, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No events occurred prior to assignment of study arm treatments.
Groups:
- 1- Leflunomide Alone - vs Combination Therapy: Group A: Leflunomide alone
  Leflunomide: A loading dose of 100 mg (or placebo) for three (3) days will be given. Following that three-day period, a dose of 20 mg/day will be maintained throughout the remainder of the study. This dose may be decreased to 10 mg/day at the discretion of the treating physician if minor toxicities occur (e.g., diarrhea, liver enzyme elevations
  Leflunomide: a loading dose of 100 mg (or placebo) for three (3) days will be given. Following that three-day period, a dose of 20 mg/day will be maintained throughout the remainder of the study. This dose may be decreased to 10 mg/day at the discretion of the treating physician if minor toxicities occur (e.g., diarrhea, liver enzyme elevations).
- Methotrexate-Sulfasalazine-Hydroxychloroquine: Methotrexate: Dose will start at 10mg/week. If total remission (according to ACR criteria) has not been achieved and labs are acceptable at the 8-week evaluation, the dosage will be increased to a dose of 15 mg/week Accordingly, if total remission has not been achieved and labs remain acceptable at the 16-week evaluation, the dosage will be increased to the top dose of 20 mg/week This dose will remain stable until the end of the study.
  Sulfasalazine: Dosing will start at 500 mg bid (1000 mg/day). This dose will remain steady until the 24-week evaluation. If total remission has not been achieved by this time and the labs remain acceptable, the dosage will be increased to the top dose of 1000 mg bid (2000 mg/day)
  Hydroxychloroquine: Dosing will be started and maintained throughout the study at a dose of 200 mg bid (400 mg/day).
  Intervention will remain as listed above.
  Methotrexate-Sulfasalazine-Hydroxychloroquine: Methotrexate:
  dosing starts at 10mg/week (4 tabs/wk
Period: Overall Study
Arm/Group | 1- Leflunomide Alone - vs Combination Therapy | Methotrexate-Sulfasalazine-Hydroxychloroquine | Leflunomide-Sulfasalazine-Hydroxychloroquine
Started | 22 | 23 | 24
Completed | 15 | 20 | 14
Not Completed | 7 | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- Leflunomide Alone - vs Combination Therapy | Methotrexate-Sulfasalazine-Hydroxychloroquine | Leflunomide-Sulfasalazine-Hydroxychloroquine | Total
Number analyzed (Participants) | 22 | 23 | 24 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 19 | 57
  >=65 years | 4 | 3 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5) | 54 (6) | 51 (4) | 52 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 16 | 45
  Male | 5 | 11 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 24 | 69

OUTCOME MEASURES:

1. Primary Outcome: Measuring the Safety and Efficacy of a New DMARD, Leflunomide Alone or in Combination With Traditional DMARD's. Participants Reaching ACR 20 Response. at 48 Weeks
Description: The combination of Methotrexate-Sulfasalazine-Hydroxychloroquine has been shown to be more effective than Methotrexate alone or the double combination of Methotrexate-Hydroxychloroquine. Primary outcome is ACR 20 response at 48 weeks.
  An ACR 20 Response is a measure of at least 20% improvement in the number of tender and swollen joints. and a 20% improvement in at least 3 of the following:
  the patient's global assessment of disease status; the patient's assessment of pain; the patient's assessment of function; the physician's global assessment of disease status; serum C-reactive protein levels.
Time Frame: 48 weeks
Population: This will result in a study power of 80%. This power has been calculated assuming an 80% efficacy of the methotrexate-sulfasalazine-hydroxychloroquine combination, an 80% efficacy of the leflunomide-sulfasalazine-hydroxychloroquine combination, and a 40% efficacy of leflunomide alone.
Measure: Count of Participants; unit: Participants
Groups:
- 1 Leflunomide Alone vs Combination Therapy: Group A: Leflunomide alone
  Leflunomide: A loading dose of 100 mg (or placebo) for three (3) days will be given. Following that three-day period, a dose of 20 mg/day will be maintained throughout the remainder of the study. This dose may be decreased to 10 mg/day at the discretion of the treating physician if minor toxicities occur (e.g., diarrhea, liver enzyme elevations
  Leflunomide: a loading dose of 100 mg (or placebo) for three (3) days will be given. Following that three-day period, a dose of 20 mg/day will be maintained throughout the remainder of the study. This dose may be decreased to 10 mg/day at the discretion of the treating physician if minor toxicities occur (e.g., diarrhea, liver enzyme elevations).
- Methotrexate-Sulfasalazine-Hydroxychloroquine: Methotrexate: start 10mg/wk. If total remission (ACR criteria) not achieved, labs acceptable at 8-wks, dose will increase to 15 mg/wk. If total remission not achieved, labs acceptable at16-wks, dose will increase to 20 mg/wk.Dose will remain stable to end of study.
  Sulfasalazine: Start at 500mg bid. Dose remain steady to 24-wks. If total remission not achieved and labs acceptable, dose to increase to 1000 mg bid.
  Hydroxychloroquine: Started and maintain throughout study at 200mg bid Intervention will as listed above.
  Methotrexate-Sulfasalazine-Hydroxychloroquine: Methotrexate:
  dosing starts at 10mg/week (4 tabs/wk). If total remission (according to ACR criteria found in Appendix II) has not been achieved and the labs are acceptable at the 8-week evaluation, the dose increased to 15 mg/week (6 tabs/wk);at the 16-week evaluation, the dose increased to 20 mg/week (8 tabs/wk). This dose will remain stable until the end of the study.
  Sulfasalazine: dosing will start at 5
Arm/Group | 1 Leflunomide Alone vs Combination Therapy | Methotrexate-Sulfasalazine-Hydroxychloroquine | Leflunomide-Sulfasalazine-Hydroxychloroquine
Number analyzed (Participants) | 22 | 23 | 24
Participants | 8 | 20 | 12

ADVERSE EVENTS:
Groups:
- Methotrexate-Sulfasalazine-Hydroxychloroquine: Methotrexate: start 10mg/wk. If remission (ACR criteria) not achieved, labs acceptable at 8-wks, dose will to 15 mg/wk. If remission not achieved, labs acceptable at16-wk, increase to 20 mg/wk.Dose stable to end of study.
  Sulfasalazine: Start at 500mg bid. Dose steady to 24-wks. If total remission not achieved/labs acceptable, dose to 1000mg bid.
  Hydroxychloroquine: Start/maintain throughout study at 200mg bid Intervention will as listed above.
  Methotrexate-Sulfasalazine-Hydroxychloroquine: Methotrexate:
  starts 10mg/wk. If total remission (according to ACR criteria) not achieved labs are acceptable at 8-wks, dose increase to 15mg/wk; at 16-wks, dose increase to 20mg/wk. Dose stable until the end of study.
  Sulfasalazine: start at 500mg bid. Dose steady to 24-wks. If total remission not achieved by this time and labs acceptable, dose will increase to 1000mg bid Hydroxychloroquine; started and maintained throughout the study at 200 mg bid
Arm/Group | 1 Leflunomide Alone vs Combination Therapy | Methotrexate-Sulfasalazine-Hydroxychloroquine | Leflunomide-Sulfasalazine-Hydroxychloroquine
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 1/22 | 2/23 | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Leflunomide Alone vs Combination Therapy (N=22) | Methotrexate-Sulfasalazine-Hydroxychloroquine (N=23) | Leflunomide-Sulfasalazine-Hydroxychloroquine (N=24)
lung carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — It was felt lung cancer was probably a result of her long smoking history; however, as she required hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Leflunomide Alone vs Combination Therapy (N=22) | Methotrexate-Sulfasalazine-Hydroxychloroquine (N=23) | Leflunomide-Sulfasalazine-Hydroxychloroquine (N=24)
GI distress (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No